CLINICAL TRIAL: NCT07315568
Title: COUPLES AND MICROBIAL DIVERSITY
Acronym: CLARITY
Status: Not yet recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R23082
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Infertility; Transmission; Infections
Keywords: Human Microbiome; HPV; Infertility; Microbial Diversity
MeSH Terms: conditions — Infertility; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will take swab samples from the cervix/vagina/anus (women), additionally penile shaft (men) as well as saliva samples and gargle samples from oral cavity from all participating. The follow-up samples are self-collected samples: saliva, oral gargle, genital sample. At birth additional sample from the placenta and breast milk are collected. From the offspring the oral, genital and anus samples are collected at the hospital and at home at six months anus ja oral sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CLARITY: Couples attending the Tampere University Hospital (TAUH) infertility clinic due to problems in conceiving during the past 12 months.

SUMMARY:
Couples and Microbial Diversity (CLARITY) - study is a prospective study that investigates the risks and dynamics of different microbes and transmission among couples to optimize the prevention and control strategies as well as improvement for infertility treatments.

The study will be conducted at the Infertility Clinic of Tampere University Hospital, Tampere Finland; and will recruit 200 couples undergoing infertility investigations and treatments. Oral and genital tract samples will be collected at baseline and every six months during a two-year follow-up period. Background information will be obtained through a secure online questionnaire.

Couples who achieve pregnancy will be followed according to the CLARITY protocol until delivery, after which families will transition to the CLARITY-Baby extension study. Samples from both the newborn and parents will be collected at delivery and again at six months postpartum, accompanied by an online follow-up questionnaire completed by the parents.

DETAILED DESCRIPTION:
Couples and Microbial Diversity (CLARITY) - study is a prospective study that investigates the risks and dynamics of different microbes and transmission among couples to optimize the prevention and control strategies as well as improvement for infertility treatments.

This research proposals main aim is to explore a variety of outcomes related to HPV-infection and other microbes and to evaluate how different variables of the mucosal ecosystem impacts these outcomes.

The study has three main parts:

PART 1. Describe couples' oral and genital HPV infections prevalence jointly with the other oral and genital microbial diversity in longitudinal setting.

PART 2. Investigate the role of different microbe infections and interactions in reproductive health and pregnancy success rate among couples enrolled for infertility treatments at the clinic.

PART 3. Provide information on the mother-child and father-child microbial vertical and horizontal transmission.

Study sets: We plan to recruit to a prospective cohort study 200 couples attending the Tampere University Hospital (TAUH) infertility clinic due to problems in conceiving during the past 12 months.

Samples: At recruitment (Baseline) we will take swab samples from vulva, cervix, vagina and anus, as well as saliva samples and gargle samples from oral cavity from all participating women. From the males otherwise same oral samples are taken as from the women, apart from genital samples that will be taken from the penile shaft, and additionally a semen sample is collected. The plan of infertility treatment itself is not affected and patients are treated according to routine practice guidelines. The follow-up samples are self-collected samples at 6, 12, 18 and 24 months (saliva, oral gargle, genital sample (in men genital sample is optional). With the extended CLARITY-Baby protocol at delivery the following additional samples will be collected: a breast milk from the mother, sample form the placenta and samples from the offspring (genital, saliva and oral brush sample).

Questionnaire: Background information of different behavioral and reproductive factors is collected using web-based self-completed questionnaires from all study participants at baseline. When necessary, the background information is completed using patient files. Secondary shorter questionnaires will be done at 12 months and 24 months of the CLARITY-protocol and at 6 months follow-up visit after delivery in the CLARITY-Baby Protocol.

Biological assays include: HPV genotyping, HLA typing, metagenomic sequencing, methylation analysis, and targeted sequencing.

Statistical analysis plans will vary by study objective and will include logistic regression, generalized estimating equations (GEE), ROC curve construction, and compositional methods for microbial profiling. All analyses will be conducted using STATA (STATA Corp., TX).

Schedule The study has been approved by the Wellbeing Services County of Pirkanmaa District Ethical Review Board. Recruitment will start in Janyary 2026.

Findings will support the development of prevention strategies, improved risk stratification, and innovative diagnostic and therapeutic approaches for couples to optimize the prevention and control strategies as well as improvement for infertility treatments.

ELIGIBILITY:
Inclusion Criteria:

* Problems in conceiving the past 12 months
* Over 18 years old
* Fluent in Finnish

Exclusion Criteria:

* Needs for donated gametes (except for female homosexual couples)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Couples attending the Tampere University Hospital (TAUH) infertility clinic due to problems in conceiving during the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Risks and dynamics of different microbes and transmission among infertile couples | From enrolment to 24 month follow-up samples
  Oral and genital samples are sequenced for various microbes with metagenomic sequencing to detect various viral, bacterial and mycobiome infections

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Louvanto, Professor, Principal Investigator — Tampere University

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Time Frame: Beginning 3 months after publication with no end date
Access Criteria: IPD that underlie the results reported in a publication, after de-identification, will be available for researchers who provide a methodologically sound proposal with achievable aims. Proposals should be directed via e-mail to the PI of the study (KL); data requestors will need to sign a data access agreement.